CLINICAL TRIAL: NCT01840748
Title: Development and Prevention of Pulmonary Hypertension in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: European Union (Other); University of Giessen (Other); University of Zurich (Other); University of Florence (Other); University of Campania Luigi Vanvitelli (Other); University of Basel (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University of Pecs (Other); University of Leeds (Other); Schoen Klinik Hamburg Eilbek (Other)
Responsible Party: Principal Investigator, Yannick ALLANORE, Prof. Yannik Allanore, University of Paris 5 - Rene Descartes
Other Study IDs: HEALTH-F5-2012-305495-OT4
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Sclerosis; Pulmonary Hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- no vasodilator: patients receiving no vasodilator
- CCB: patients receiving a calcium channel blocker (CCB) for digital vasculopathy
- i.v. prostanoids or PDE5i or ETRAs: patients treated with i.v. prostanoids or phosphodiesterase-5 inhibitors (PDE5i) or endothelin receptor antagonists (ETRA), regardless of whether a calcium channel blocker is given in addition

SUMMARY:
Systemic sclerosis (SSc) is an orphan, multiorgan disease affecting the connective tissue of the skin and several internal organs.

Pulmonary hypertension (PH) is a fatal disorder characterized by an increase in pulmonary vascular resistance, which leads to right ventricular failure. Despite being recently the object of greater attention and despite therapeutic advances, pulmonary hypertension due to SSc remains associated with a dismal 47 - 67% 3-year survival. Among SSc patients prospectively followed in the "European League Against Rheumatism Scleroderma Trials and Research" (EUSTAR) cohort, 26% of death was related to pulmonary hypertension. Although some previous data have suggested the protective effects of calcium channel blockers on the development of pulmonary hypertension, the potential preventive effects of vasodilators for the prevention of Pulmonary hypertension have not been determined yet. In addition to be considered routinely for the treatment of SSc-related pulmonary hypertension, prostanoids, endothelin receptor antagonists (ETRA) and Phosphodiesterase-5 inhibitors (PDE5i) can also be used for this indication.

This observational trial is one out of five observational trials of the collaborative project "To decipher the optimal management of systemic sclerosis" (DeSScipher).

Aim of this observational trial is:

- to compare the outcomes of adult and juvenile SSc patients who are at high risk of developing pulmonary hypertension and are receiving either different vasodilator treatments or no vasodilator treatment.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile and adult Systemic sclerosis patients, with diagnosis according to the ACR/EULAR adult SSc criteria and PRES/ACR/EULAR juvenile SSc criteria respectively
* Patients at high risk of pulmonary hypertension with a Cochin Risk prediction score >/= 3

ACR = American College of Rheumatology; EULAR = European League Against Rheumatism; PRES = Pediatric Rheumatology European Society

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are adult and juvenile systemic sclerosis patients from the EUSTAR cohort (MEDSonline database) and the juvenile systemic sclerosis working group cohort
Sampling Method: Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The number of patients with pulmonary hypertension at 2 years | 2 years

SECONDARY OUTCOMES:
Time to development of precapillary pulmonary hypertension | 2 years
  participants will be followed for the duration of 2 years, the time until development of precapillary pulmonary hypertension is the secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Allanore, Prof., Principal Investigator — Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016; Ulf Müller-Ladner, Prof., Study Chair — Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology
Locations (11):
- Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016, Paris, France
- Germany (3):
  - Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Centre for Pediatric Rheumatology, Klinikum Eilbek, Hamburg
- Pecsi Tudomanyegyetem - University of Pecs, Pécs, Hungary
- Italy (2):
  - University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine, Florence
  - Policlinico, Via Pansini, Napoli-Italia
- Switzerland (2):
  - Felix-Platter Spital, University of Basel, Basel
  - University of Zurich, Department of Rheumatology, Zurich
- United Kingdom (2):
  - The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital, Leeds
  - Royal Free Hospital, University College London, London